CLINICAL TRIAL: NCT00762086
Title: A Prospective, Randomized, Multi-center Clinical Trial to Evaluate the Efficacy and Safety of a New Intermittent Pneumatic Compression Device on Initial Claudication Distance in Patients With Peripheral Arterial Disease Stage II.
Brief Title: Safety and Efficacy Study of a New Intermittent Pneumatic Compression Device to Treat Patients With Peripheral Arterial Disease (PAD) Stage II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mego Afek Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HM-AHR-01
Record Dates: First submitted 2008-09-28; First posted 2008-09-30 (Estimated); Results first posted 2012-08-27 (Estimated); Last update posted 2012-08-31 (Estimated); Status verified 2012-08

CONDITIONS: Peripheral Arterial Disease
Keywords: Peripheral Arterial Disease; intermittent pneumatic compression treatment; Initial claudication
MeSH Terms: conditions — Peripheral Arterial Disease | interventions — Dosage Forms

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment Group (Active Comparator): AngioPress Intermittent pneumatic compression (IPC) Device
  Interventions: Device: AngioPress Intermittent pneumatic compression (IPC) Device
- Control Group (Other): Aspirin/Clopidegrol and Standard walking exercises
  Interventions: Other: Medications and Standard walking exercises

INTERVENTIONS:
Device: AngioPress Intermittent pneumatic compression (IPC) Device — Treatment with Intermittent pneumatic compression (IPC) for PAD
  Arms: Treatment Group
Other: Medications and Standard walking exercises — Aspirin/Clopidegrol and Standard walking exercises
  Arms: Control Group

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of new intermittent pneumatic compression device on initial claudication distance in patients with Peripheral Arterial Disease stage II

DETAILED DESCRIPTION:
Patients with Peripheral Arterial Disease (PAD) suffer from symptoms such as intermittent claudication, limb and foot pain and tissue lesions, which are difficult to treat. In recent years, there have been reports demonstrating reduction of these symptoms by use of compressible sleeve devices.

This clinical study aims at demonstrating the safety and effectiveness of this device in treating PAD symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subject 18 to 90 years, of any race.
* Patients with proven Peripheral Arterial Disease (PAD) in Doppler Ultrasound and Ankle-Brachial Pressure Index (ABPI ≤ 0.9 in one leg)
* Subject with stable (>3 month) PAD Fontaine Stage II.
* Aortoiliac vessels with no significant hemodynamic disturbances , as confirmed by recent (<30 days) clinical examination
* Subject has intermittent claudication and claudication pain of the calf
* Subject has stable intermittent claudication (>3 month and not more than one year) with initial claudication distance not more than 250 meters, as determined by treadmill test (3.2 km/h, 10% grade)
* Subject willing to participate as evidenced by signing the written informed consent.
* Treatment with Aspirin or Clopidogrel for at least 7 days
* Willingness to undergo standardized walking exercise

Exclusion Criteria:

* Ankle-Brachial Pressure Index (ABI) above 0.8 in both legs. In Diabetic patients with no compressible arteries ABI above 40 mm/Hg of the higher pressure measured in both arms.
* Inability to walk
* Chronic respiratory insufficiency (severe obstructive or restrictive)
* Coronary artery disease with angina
* Stroke, myocardial infarction or other acute vascular events in the last 3 months
* Mild-Severe congestive heart failure
* Degenerative or inflammatory hip, knee, ankle or foot joint lesions interfering with walking
* Spinal stenosis or disc lesions with lower limb motor sensory defects
* Leg trauma, limb or skin infection or edema
* Recent (6 months) abdominal, cardiothoracic, vascular or orthopedic (lower limb) surgery
* Subject after crural or pedal bypass surgery
* Subject with neuropathy
* Uncontrolled arterial hypertension
* Morbid obesity (BMI >35.0)
* Need for concomitant medication with potential vascular activity
* Routinely use of pain relief medications (i.e. NSAIDs, Narcotics etc)
* Expected weak compliance
* Subject requires surgical or endovascular intervention for PAD
* Subject has known allergy to device components (sleeve fabric).
* Subject has medical conditions that may be worsened by concomitant use of the device (i.e. recent (1 year) Deep Vein Thrombosis).
* Subject participates in any other clinical study at the same time

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2009-03; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Avigdor Zelikovski, Prof., Principal Investigator
Locations (4):
- Germany (2):
  - Praxis für Angiology, Munich
  - Praxis für Gefäßmedizin am Tegernsee, Rottach-Egern
- Israel (2):
  - Bnai Zion Medical Center, Haifa
  - NARA Medical Center, Ramat Gan

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between March 2009 and August 2011, a total of 67 patients were screened and randomized into the study. Patients were recruited from private clinics and clinics affiliated to University Hospitals
Pre-assignment Details: Subjects were required to be treated with Aspirin/Clopidogrel for at least one week priot to 1st treatment
Groups:
- Treatment Group: AngioPress IPC Device
Period: Overall Study
Arm/Group | Treatment Group | Control Group
Started | 39 | 28
Completed | 33 | 24
Not Completed | 6 | 4
Not completed — Adverse Event | 2 | 0
Not completed — Lost to Follow-up | 0 | 2
Not completed — Non compliance | 1 | 0
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Ineligible to participate in the study | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Group | Control Group | Total
Number analyzed (Participants) | 39 | 28 | 67
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 11 | 22
  >=65 years | 28 | 17 | 45
Age Continuous [Mean (Standard Deviation); unit: years] | 70.8 (6.96) | 67.8 (11.76) | 69.5 (9.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 5 | 17
  Male | 27 | 23 | 50
Region of Enrollment [Number; unit: participants]
  Israel | 25 | 23 | 48
  Germany | 14 | 5 | 19

OUTCOME MEASURES:

1. Primary Outcome: Absolute Claudication Distance (ACD)
Description: Absolute walking distance is measured by walking on a treadmill until the point when the subject is inable to walk anymore due to pain in the leg. The walking distance is measured by meters
Time Frame: 3 months
Population: ITT cohort
Measure: Least Squares Mean (Standard Error); unit: Meters
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 39 | 28
Meters | 54.374 (15.3752) | 0.792 (18.0868)

ADVERSE EVENTS:
Arm/Group | Treatment Group | Control Group
Serious Adverse Events (participants affected / at risk) | 2/39 | 0/28
Other Adverse Events (participants affected / at risk) | 2/39 | 0/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Group (N=39) | Control Group (N=28)
Hypertensive Crisis (Cardiac disorders) | 1 (1) | 0 (0)
Congestive heart failure (Cardiac disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Group (N=39) | Control Group (N=28)
Application site discomfort (General disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No